CLINICAL TRIAL: NCT03141385
Title: Renal Effects of Remote Ischemic Preconditioning in Patients After Total Arch Replacement
Brief Title: Renal Effects of RIPC in Patients After Total Arch Replacement
Acronym: RenRIPC-TAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Guyan Wang, The Chief of Infection-Control Department, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FW2016-F09
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Acute Kidney Injury; Dialysis
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIPC intervention (Experimental): Remote ischemic preconditioning (RIPC) will be induced after the general anesthesia prior to the cardiopulmonary bypass by four cycles of right limber ischemia (5-min blood pressure cuff inflation to a pressure of 200mmHg or a pressure that is 50 mmHg higher than SAP and 5-min cuff deflation)
  Interventions: Other: remote ischemic preconditioning
- Control (Sham Comparator): Four cycles of right upper limb pseudo ischemia and reperfusion, which will be induced by 5-minute blood pressure cuff inflation to a low pressure of 20 mmHg followed by 5-minute cuff deflated.
  Interventions: Other: Control

INTERVENTIONS:
Other: remote ischemic preconditioning — Remote ischemic preconditioning (RIPC) will be induced after the general anesthesia prior to the cardiopulmonary bypass by four cycles of right limber ischemia (5-min blood pressure cuff inflation to a pressure of 200mmHg or a pressure that is 50 mmHg higher than SAP and 5-min cuff deflation)
  Arms: RIPC intervention
Other: Control — Four cycles of right upper limb pseudo ischemia and reperfusion, which will be induced by 5-minute blood pressure cuff inflation to a low pressure of 20 mmHg followed by 5-minute cuff deflated.
  Arms: Control

SUMMARY:
The purpose of this study is to test the hypothesis that remote ischemic preconditioning prevents acute kidney injury and improves clinical outcomes in patients undergoing total arch replacement.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a well-recognized complication after cardio-thoracic surgeries and is associated with increased morbidity and mortality. Total arch replacement is reported with a relatively high incidence of post-operative AKI. In addition, few effective preventive or therapeutic interventions for AKI have been identified. A number of studies have now addressed renal protection as a primary outcome following RIPC. Because the mechanism of I/R injury are similar to those proposed for AKI after CPB, the purpose of this study is to test the hypothesis that remote ischemic preconditioning prevents acute kidney injury and improves clinical outcomes in patients undergoing total arch replacement.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for total arch replacement
* written informed consent

Exclusion Criteria:

* pre-existing AKI
* peripheral vascular disease affecting the upper limbs
* hybrid total arch replacement
* the history of kidney transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence of AKI within the 7 days after the surgery | Within 7 days after the surgery
  AKI defined by KDIGO criteria

SECONDARY OUTCOMES:
Incidence of severe AKI (stage 2 and stage 3) | Within 7 days after the surgery
  severity defined by KDIGO criteria
Renal replacement therapy | Within 30 days after the surgery
  the requirement for RRT during index hospital stay
Mechanical ventilation duration | Within 30 days after the surgery
  duration of mechanical ventilation in the intensive care unit
Length of intensive care unit stay | Within 30 days after the surgery
  length of stay on the intensive care unit
In-hospital death | Within 30 days after the surgery
  in-hospital all-cause death
Stroke | Within 30 days after the surgery
  new onset stroke during index hospital stay
Paraplegia | Within 30 days after the surgery
  impairment in motor or sensory function of the lower extremities during index hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Guyan Wang, PhD, Principal Investigator — State Key Laboratory of Cardiovascular Disease, Fuwai Hospital, National Center for Cardiovascular Diseases, CAMS and PUMC, Beijing, China
Locations (1):
- State Key Laboratory of Cardiovascular Disease, Fuwai Hospital, National Center for Cardiovascular Diseases, CAMS and PUMC, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250
- [Derived] Chen Y, Wang G, Zhou H, Yang L, Zhang C, Yang X, Lei G. 90 days impacts of remote ischemic preconditioning on patients undergoing open total aortic arch replacement: a post-hoc analysis of previous trial. BMC Anesthesiol. 2020 Jul 9;20(1):169. doi: 10.1186/s12871-020-01085-9. PMID 32646379
- [Derived] Zhou H, Yang L, Wang G, Zhang C, Fang Z, Lei G, Shi S, Li J. Remote Ischemic Preconditioning Prevents Postoperative Acute Kidney Injury After Open Total Aortic Arch Replacement: A Double-Blind, Randomized, Sham-Controlled Trial. Anesth Analg. 2019 Jul;129(1):287-293. doi: 10.1213/ANE.0000000000004127. PMID 30896603